CLINICAL TRIAL: NCT00821990
Title: A Patient Preference Randomized Phase III Clinical Trial of Second-line Chemotherapy (SLC) in Advanced Gastric Cancer (AGC) Patients Pretreated With Both Fluoropyrimidines and Platinum
Brief Title: Second-line Therapy Versus Supportive Care for Pretreated Advanced Gastric Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Se Hoon Park, MD, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-08-055
Record Dates: First submitted 2008-12-29; First posted 2009-01-14 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Failed after previous chemotherapy
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chemotherapy (Active Comparator): Eligible patients will be first offered randomization. If willing to participate RCT, the patient will be randomized to chemotherapy or best supportive care. If patients refuse to participate in RCT, but nevertheless agree to receive treatment of their preferences, they are offered their treatment of choice (chemotherapy or supportive care).
  Interventions: Drug: Chemotherapy; Other: Best supportive care
- Supportive care (Active Comparator): Eligible patients will be first offered randomization. If willing to participate RCT, the patient will be randomized to chemotherapy or best supportive care. If patients refuse to participate in RCT, but nevertheless agree to receive treatment of their preferences, they are offered their treatment of choice (chemotherapy or supportive care).
  Interventions: Other: Best supportive care

INTERVENTIONS:
Drug: Chemotherapy — The administration of chemotherapy regimen (docetaxel or irinotecan) will be determined at the discretion of investigator, and depends on the patient's previous chemotherapy.
  Arms: Chemotherapy
Other: Best supportive care — It includes nutritional support, analgesics, antibiotics, antiemetics, transfusions, or any other symptomatic therapy (with the exception of cytotoxic chemotherapy) and/or assistance of a psychological support. Localized radiotherapy to alleviate symptoms such as pain is allowed provided that the total dose delivered is in a palliative range.

SUMMARY:
Because well-designed, randomized, controlled clinical trials are lacking in patients with advanced gastric cancer (AGC), and because randomly allocating patients to treatments that do not accord with their preferences may influence trial validity, the investigators employed a patient preference randomized trial design to compare the efficacy of second-line chemotherapy and best supportive care.

DETAILED DESCRIPTION:
Fluoropyrimidine and/or platinum-based chemotherapy is now regarded as a standard first-line treatment in AGC patients because it has shown superiority in terms of response rate and time to disease progression compared with 5-FU monotherapy and other combinations in phase III trials. Despite the lack of evidence for benefit associated with administering salvage chemotherapy, it is a common practice to offer further chemotherapy for AGC patients after first-line failure. For patients who failed after fluoropyrimidine and platinum, taxanes (paclitaxel or docetaxel) and irinotecan have been evaluated extensively in the second-line setting.

Currently, there is no evidence that SLC in patients with AGC will result in substantial prolongation of survival and there is potential for toxicity from the treatment.

ELIGIBILITY:
Inclusion Criteria:

* aged 75 year or younger
* advanced gastric cancer
* ECOG performance status 0 or 1
* previous failure after chemotherapy with fluoropyrimidine and platinum
* adequate major organ functions

Exclusion Criteria:

* severe concurrent illness and/or active infection
* previously treated with taxanes and irinotecan
* active CNS metastases
* pregnant or lactating women
* who have not recovered from prior treatments

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Survival | 1 year after last patient entered

CONTACTS AND LOCATIONS:
Overall Officials: Se Hoon Park, MD, Principal Investigator — Samsung Medical Center, Seoul, Korea
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Wagner AD, Grothe W, Haerting J, Kleber G, Grothey A, Fleig WE. Chemotherapy in advanced gastric cancer: a systematic review and meta-analysis based on aggregate data. J Clin Oncol. 2006 Jun 20;24(18):2903-9. doi: 10.1200/JCO.2005.05.0245. PMID 16782930
- [Background] Wilson D, Hiller L, Geh JI. Review of second-line chemotherapy for advanced gastric adenocarcinoma. Clin Oncol (R Coll Radiol). 2005 Apr;17(2):81-90. doi: 10.1016/j.clon.2004.10.006. PMID 15830569